CLINICAL TRIAL: NCT01850836
Title: Treatment of Aphasic Stroke Patients With rTMS
Brief Title: Dual Hemisphere rTMS for Rehabilitation of Post Stroke Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman M. Khedr, Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: rTMS in Rehab of aphasia
Record Dates: First submitted 2013-03-12; First posted 2013-05-10 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2013-05

CONDITIONS: Non Fluent Aphasia in Subacute Stroke
Keywords: Aphasia, Stroke, repetitive transcranial magnetic stimulation.
MeSH Terms: conditions — Aphasia; Stroke | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Real rTMS (Active Comparator): 19 subacute stroke pts with aphasia received 10 rTMS (5sessions/week) for 2 successive weeks
  Interventions: Procedure: repetitive transcranial magnetic stimulation
- Sham rTMS (Sham Comparator): 10 patients received sham rTMS stimulation (5 sessions/week) for 2 successive weeks
  Interventions: Procedure: repetitive transcranial magnetic stimulation

INTERVENTIONS:
Procedure: repetitive transcranial magnetic stimulation
  Other Names: rTMS

SUMMARY:
To investigate the therapeutic effect of dual hemisphere repetitive transcranial magnetic stimulation (rTMS) on post-stroke non fluent aphasia.

DETAILED DESCRIPTION:
Thirty patients with subacute post-stroke non-fluent aphasia were randomly allocated with a ratio 2:1 to receive real (n = 20) or sham (n = 10) rTMS of the affected motor cortex. Each patient received 1000 rTMS pulses (1 Hertz at 110% of resting motor threshold) over the unaffected Broca's area and 1000 pulses (20 Hertz at 100% resting motor threshold) over affected left Broca's area for 10 consecutive days. LANGUAGE section of hemispheric stroke scale, Stroke Aphasic Depression Questionnaire Hospital Version (SADQ-H) and NIH stroke scale were assessed before, post sessions, 1 and 2 months after the last session . Motor threshold was assessed before and after the end of last session.

ELIGIBILITY:
Inclusion Criteria:

* acute hemiplegia with non-fluent aphasia, single thromboembolic non-haemorrhagic infarction documented by computerized tomography (CT) in the distribution of middle cerebral artery.

Exclusion Criteria:

* head injury or neurological disease other than stroke,
* Unstable cardiac dysrhythmia,
* Fever,
* Infection,
* Hyperglycaemia
* Prior administration of tranquilizer
* Patients with no motor evoked response recorded from first dorsal interosseus (FDI) muscle of the affected hand

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-12; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Hemispheric stroke scale (HSS) | Change from Baseline in HSS at 2 months
  Language assessment using hemispheric stroke scale (HSS)

SECONDARY OUTCOMES:
NIH Stroke Scale (NIHSS) | Change from Baseline in NIHSS at 2 months

OTHER OUTCOMES:
Stroke Aphasic Depression Questionnaire Hospital Version (SADQ-H) | Change from Baseline in SADQ-H at 2 months
  (Asking about presence of depressive symptoms within last week of stroke to be present all the days or frequent from 4-6 days, or infrequent from 1-4 days, or not at all).